CLINICAL TRIAL: NCT05912205
Title: An Open, Single Arm, Phase II Clinical Study on the Efficacy and Safety of Bladder Sparing Therapy With Vidixizumab Combined With Local Radiotherapy in Patients With HER-2 Expressing Myometrial Invasive Urothelium Carcinoma
Brief Title: Disitamab Vedotin Combined With Radiotherapy for Bladder Preservation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT221037
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — disitamab vedotin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin combined with radiotherapy (Experimental): Disitamab Vedotin (RC48) 2.0mg/kg, once every two weeks, intravenous drip (60-90 min); Radiotherapy (SBRT, bladder irradiation field with a total dose greater than 50 Gy)
  Interventions: Drug: Disitamab Vedotin; Radiation: radiotherapy

INTERVENTIONS:
Drug: Disitamab Vedotin — Four cycles of neoadjuvant therapy with Vidiximab (2.0mg/kg) were administered first, followed by bladder sparing therapy using maximized TURBT combined with radiotherapy and chemotherapy. The patient will receive vidiximab combined with local radiotherapy after maximizing TURBT surgery. The subjects received treatment with Vidixitol every two weeks for six consecutive treatment cycles, and simultaneously received 1 month of radiation therapy (SBRT, total dose of bladder irradiation field greater than 50 Gy)
Radiation: radiotherapy — radiotherapy

SUMMARY:
This is a prospective, open, single center clinical study of vidicizumab combined with local radiotherapy as bladder conserving therapy in patients with muscle invasive bladder urothelium cancer with HER-2 expression (IHC 2+or 3+). A total of 30 subjects were included in the study

DETAILED DESCRIPTION:
A total of 30 subjects were included in the study. Each subject underwent diagnostic bladder resection (TURBT) and imaging diagnosis, and biological samples such as blood, urine, and biopsy tissue were collected before treatment. After myometrial invasive bladder cancer with HER2 expression (IHC 2+or 3+) judged by pathological tissue, four cycles of neoadjuvant therapy with vedixizumab (2.0mg/kg) was first performed, and then bladder conserving therapy was performed by maximizing TURBT combined with radiotherapy and chemotherapy. The patient will receive vidiximab combined with local radiotherapy after maximizing TURBT surgery. The subjects received a treatment cycle of six consecutive treatment cycles of vidixitol every two weeks, and simultaneously received one month of radiation therapy (SBRT, with a total dose of over 50 Gy in the bladder irradiation field). After completing the above treatment, tumor evaluation will be conducted through imaging and exfoliative cytology. After the completion of radiotherapy, the first tumor efficacy evaluation will be conducted. After the end of radiotherapy, tumor efficacy evaluation will be conducted every 6 weeks. Patients who are not tolerant to radiotherapy (evaluated by the researchers) will directly discontinue the medication.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years old;
2. ECOG PS: 0-1 points;
3. Subjects need to receive cystoscope or diagnostic electrotomy, imaging diagnosis, and the investigator judges that it is myometrial invasive bladder urothelium cancer (urothelium cancer is the main pathological component>50%), and plans to receive comprehensive treatment for bladder preservation;
4. Clinical staging T2 (CT/MRI+PET/CT);
5. Expected survival time ≥ 3 months;
6. The immunohistochemical staining result of the tissue after cystoscope or diagnostic electrotomy was IHC 2+or 3+;
7. The main organ function is normal (14 days before enrollment), which meets the following criteria:

(1) The blood routine examination standard should meet (no blood transfusion or granulocyte colony-stimulating factor treatment within 14 days before enrollment): HB ≥ 90 g/L; ANC ≥ 1.5 × 109/L; PLT ≥ 100 × 109/L; 8. Have not received systemic corticosteroid therapy within 4 weeks prior to treatment; 9. Men with reproductive ability or women with the possibility of pregnancy must use highly effective contraceptive methods during the trial process and continue to use contraception for 12 months after the end of treatment; 10. The subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Those who have received other anti-tumor treatments (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks prior to the start of research treatment, or have not yet recovered from previous toxicity (excluding 2 degree hair loss and 1 degree neurotoxicity
2. Pregnant or lactating women;
3. Positive HIV test results;
4. Active hepatitis B or C patients
5. Have a clear history of active tuberculosis;
6. Active autoimmune diseases that require systematic treatment within the past 2 years (such as the use of disease regulating drugs, corticosteroids, or immunosuppressive drugs), allowing relevant alternative treatments (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for renal or pituitary dysfunction);
7. Other serious and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results.
8. Urothelium carcinoma of upper urinary tract (urothelium carcinoma of renal pelvis and ureter)
9. According to the researcher's perspective, there may be increased risks associated with participating in the study, or other severe, acute, or chronic medical or mental illnesses or laboratory abnormalities that may interfere with the interpretation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Bladder-intact event-free survival | 1 year
  1-year event free survival with intact bladder

SECONDARY OUTCOMES:
Pathologic Complete Response | 2 mouths
  Neoadjuvant therapy and postoperative pathology confirmed that the primary tumor was in complete remission (stage ypT0) and had no residual tumor cells, regardless of whether the regional lymph nodes were involved or not.

CONTACTS AND LOCATIONS:
Overall Officials: zhang xiaoping, doctor, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology

IPD SHARING:
Plan to Share IPD: No
not share